CLINICAL TRIAL: NCT02759354
Title: Long-term Persistence of Hepatitis B and Pertussis Antibody Responses in Healthy 4 to 5 Year-Old Children Previously Vaccinated With a 2-Dose or 3-Dose Infants Series and Toddler Dose With Vaxelis® or INFANRIX® Hexa
Brief Title: Long-term Persistence of Hepatitis B and Pertussis Antibody Responses in Healthy 4 to 5 Year Old Children Previously Vaccinated With Vaxelis® or INFANRIX® Hexa (V419-012)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MCM Vaccines B.V. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V419-012; 2016-000274-37 (Other: EudraCT Number); PRI03C (Other: MCMVaccBV Protocol ID); V419-012 (Other: Merck Protocol Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis B; Pertussis
Keywords: Immune response
MeSH Terms: conditions — Hepatitis B; Whooping Cough | interventions — Blood Specimen Collection; Vaxelis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group Vaxelis (3+1) (Experimental): Participants previously vaccinated with a 3-dose primary series of Vaxelis® at 2, 3 and 4 months of age, and a toddler dose at 12 months of age (study V419-007).
  Interventions: Other: Blood Sample
- Group Infanrix hexa (3+1) (Active Comparator): Participants previously vaccinated with a 3-dose primary series of INFANRIX® hexa at 2, 3 and 4 months of age, and a toddler dose at 12 months of age (study V419-007).
  Interventions: Other: Blood Sample
- Group Vaxelis (2+1) (Experimental): Participants previously vaccinated with a 2-dose primary series of Vaxelis® at 2 and 4 months of age, and a toddler dose at 11-12 months of age (study V419-008).
  Interventions: Other: Blood Sample
- Group Infanrix hexa (2+1) (Active Comparator): Participants previously vaccinated with a 2-dose primary series of INFANRIX® hexa at 2 and 4 months of age, and a toddler dose at 11-12 months of age (study V419-008).
  Interventions: Other: Blood Sample

INTERVENTIONS:
Other: Blood Sample — Blood sample at approx. 4 years of age
  Other Names: Vaxelis®; INFANRIX® hexa

SUMMARY:
This is a multicenter extension study of two European randomized, double-blind studies (V419-007 and V419-008). It describes long-term persistence of hepatitis B and pertussis antibody responses in healthy 4- to 5 year old children previously vaccinated with Vaxelis® or INFANRIX® hexa

ELIGIBILITY:
Inclusion Criteria

1. Healthy child of either gender, who has received a complete 3-dose primary series or a complete 2 dose primary series followed by a toddler dose with VAXELIS or INFANRIX hexa as part of the V419-007 or V419-008 study respectively.
2. Informed consent signed by the participant's parent(s) or legal representative.

Exclusion Criteria:

1. Participant who has received any dose of hepatitis B (HB)-containing vaccine at any time other than study vaccine in V419-007 or V419-008 study.
2. Participant with a history of diagnosis (clinical, serological or microbiological) of HB virus infection of the V419-007 or V419-008 study.
3. Participant who has received any dose of pertussis-containing vaccine after completion of the V419-008 study.
4. Participant with a history of diagnosis (clinical, serological or microbiological) of infection due to pertussis after completion of V419-008 study.
5. Participation at the time of study enrolment or in the 4 weeks preceding the study enrolment in another clinical study investigating a vaccine, drug medical device, or medical procedure*.
6. Participant who received immunoglobulins, blood or blood-derived products within 3 months prior to inclusion*.
7. Receipt of immunosuppressive therapy or other immune-modifying drugs, such as anti-cancer chemotherapy or radiation therapy since completion of V419-007 or V419-008 studies.
8. Participant with suspected or known blood dyscrasias, leukemia, lymphomas of any type or other malignant neoplasms affecting the haematopietic and lymphatic systems since completion of V419-007 or V419-008 studies.

   * Criteria 5 and 6 are temporary exclusion criteria. If a participant meets criteria 5 and/or 6 at the time of Visit 1, a further appointment is to be scheduled to reassess the participant's eligibility.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 754 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Vesikari T, Xu J, Johnson DR, Hall J, Marcek T, Goveia MG, Acosta CJ, Lee AW. Hepatitis B and pertussis antibodies in 4- to 5-year-old children previously vaccinated with different hexavalent vaccines. Hum Vaccin Immunother. 2020 Apr 2;16(4):867-874. doi: 10.1080/21645515.2019.1673119. Epub 2019 Nov 5. PMID 31689166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter extension study was conducted in Finland at approximately 10 sites from studies V419-007 and V419-008, which had eligible participants(i.e. participants who completed the full 3+1 or 2+1 vaccination schedule in the original studies).
Pre-assignment Details: Of the 760 screened participants, 754 were enrolled and completed the study. A total of 752 participants were included in the Persistence Analysis Set, 752 with blood samples available for hepatitis B surface antigen (HBsAg) analyses, and 751 for pertussis analyses.
Groups:
- Group Vaxelis (3+1): Participants previously vaccinated with a 3-dose primary series of Vaxelis® at 2, 3 and 4 months of age, and a toddler dose at 12 months of age (study V419-007). On Day 1 of this extension study (~4 years after completion of the 3+1 schedule), a 4 mL blood sample was obtained to assay for long-term antibody persistence.
- Group Infanrix Hexa (3+1): Participants previously vaccinated with a 3-dose primary series of INFANRIX® hexa at 2, 3 and 4 months of age, and a toddler dose at 12 months of age (study V419-007). On Day 1 of this extension study (~4 years after completion of the 3+1 schedule), a 4 mL blood sample was obtained to assay for long-term antibody persistence.
- Group Vaxelis (2+1): Participants previously vaccinated with a 2-dose primary series of Vaxelis® at 2 and 4 months of age, and a toddler dose at 11-12 months of age (study V419-008). On Day 1 of this extension study (~4 years after completion of the 2+1 schedule), a 4 mL blood sample was obtained to assay for long-term antibody persistence.
- Group Infanrix Hexa (2+1): Participants previously vaccinated with a 2-dose primary series of INFANRIX® hexa at 2 and 4 months of age, and a toddler dose at 11-12 months of age (study V419-008). On Day 1 of this extension study (~4 years after completion of the 2+1 schedule), a 4 mL blood sample was obtained to assay for long-term antibody persistence.
Period: Overall Study
Arm/Group | Group Vaxelis (3+1) | Group Infanrix Hexa (3+1) | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Started | 192 | 190 | 181 | 191
Completed | 192 | 190 | 181 | 191
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants previously vaccinated in studies V419-007 or V419-008 and with immunogenicity results available were included in the Persistence Analysis Set. 754 participants completed the study but only 752 were included in the Persistence Analysis Set (2 participants had protocol deviations).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Vaxelis (3+1) | Group Infanrix Hexa (3+1) | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1) | Total
Number analyzed (Participants) | 191 | 189 | 181 | 191 | 752
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.8 (0.2) | 4.8 (0.2) | 3.9 (0.1) | 3.9 (0.1) | 4.4 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 86 | 84 | 94 | 362
  Male | 93 | 103 | 97 | 97 | 390

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Responding to Hepatitis B Surface Antigen (HBsAg)
Description: Participant serum samples were collected for testing with an enhanced chemiluminescence assay for antibodies to HBsAg. Response was defined as a titer >=10 milli International units (mIU)/mL. Confidence Intervals were calculated based on the exact binomial method of D. Collett.
Time Frame: Day 1 (approximately 4 years after completion of the 3+1/2+1 schedule)
Population: All analyses were performed on the Persistence Analysis Set, defined as all participants previously vaccinated (with a complete 3+1 or 2+1 schedule, as part of studies V419-007 or V419-008) with available immunogenicity data for the respective endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group Vaxelis (3+1) | Group Infanrix Hexa (3+1) | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 191 | 189 | 181 | 190
Percentage of Participants | 70.16 [63.13 to 76.55] | 82.01 [75.78 to 87.21] | 65.75 [58.34 to 72.63] | 83.68 [77.65 to 88.64]

2. Secondary Outcome: Geometric Mean Concentration of Antibodies to HBsAg
Description: Participant serum samples were collected for testing with an enhanced chemiluminescence assay for antibodies to HBsAg. The unit of measure is milli International Units/mL (mIU/mL). Confidence Intervals were calculated based on the t-distribution of the log-transformed antibody concentration.
Time Frame: Day 1 (approximately 4 years after completion of the 3+1 or 2+1 schedule)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Group Vaxelis (3+1) | Group Infanrix Hexa (3+1) | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 191 | 189 | 181 | 190
mIU/mL | 24.43 [19.52 to 30.59] | 51.30 [40.19 to 65.46] | 19.44 [15.48 to 24.40] | 71.00 [54.94 to 91.77]

3. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin. The unit of measure is ELISA units/mL (EU/mL). Confidence Intervals were calculated based on the t-distribution of the log-transformed antibody concentration.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: The analysis population was the Persistence Analysis Set, all participants previously vaccinated with complete 2+1 schedule (V419-008) with available immunogenicity data for the respective endpoint. Due to pre-school enrollment and booster administration, assessment of pertussis antibody persistence was not possible for the 3+1 schedule (V419-007).
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 178 | 188
EU/mL | 5.31 [4.61 to 6.12] | 3.64 [3.24 to 4.09]

4. Primary Outcome: Percentage of Participants Responding to Pertussis Toxin
Description: Participant serum samples were collected for testing with an Enzyme-linked Immunosorbent Assay (ELISA) for antibodies to pertussis toxin. The unit of measure is ELISA units/mL. The lower limit of quantification (LLOQ)=4 EU/mL. Confidence Intervals were calculated based on the exact binomial method of D. Collett.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 178 | 188
Percentage of participants
  Concentration ≥LLOQ | 58.43 [50.82 to 65.75] | 41.49 [34.37 to 48.89]
  Concentration ≥2×LLOQ | 40.45 [33.17 to 48.05] | 21.81 [16.13 to 28.40]
  Concentration ≥4×LLOQ | 14.61 [9.77 to 20.67] | 3.72 [1.51 to 7.52]

5. Primary Outcome: Percentage of Participants Responding to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin. LLOQ=3 EU/mL. Confidence Intervals were calculated based on the exact binomial method of D. Collett.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 173 | 188
Percentage of participants
  Concentration ≥LLOQ | 80.92 [74.27 to 86.49] | 88.30 [82.82 to 92.52]
  Concentration ≥2×LLOQ | 46.82 [39.21 to 54.54] | 70.74 [63.68 to 77.14]
  Concentration ≥4×LLOQ | 26.01 [19.65 to 33.22] | 45.21 [37.96 to 52.62]

6. Primary Outcome: Percentage of Participants Responding to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin. LLOQ=4 EU/mL. Confidence Intervals were calculated based on the exact binomial method of D. Collett.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 180 | 190
Percentage of participants
  Concentration ≥LLOQ | 66.11 [58.70 to 72.99] | 72.63 [65.71 to 78.84]
  Concentration ≥2×LLOQ | 43.89 [36.52 to 51.47] | 51.05 [43.71 to 58.36]
  Concentration ≥4×LLOQ | 15.56 [10.59 to 21.69] | 18.42 [13.18 to 24.68]

7. Primary Outcome: Percentage of Participants Responding to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae. LLOQ=4 EU/mL. Confidence Intervals were calculated based on the exact binomial method of D. Collett.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 177 | 183
Percentage of participants
  Concentration ≥LLOQ | 94.35 [89.86 to 97.26] | 3.28 [1.21 to 7.00]
  Concentration ≥2×LLOQ | 88.14 [82.44 to 92.50] | 2.19 [0.60 to 5.50]
  Concentration ≥4×LLOQ | 69.49 [62.14 to 76.18] | 1.09 [0.13 to 3.89]

8. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin. Confidence Intervals were calculated based on the t-distribution of the log-transformed antibody concentration.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 173 | 188
EU/mL | 6.62 [5.54 to 7.91] | 11.05 [9.13 to 13.37]

9. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin. Confidence Intervals were calculated based on the t-distribution of the log-transformed antibody concentration.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 180 | 190
EU/mL | 5.94 [5.14 to 6.86] | 7.19 [6.20 to 8.33]

10. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae. Confidence Intervals were calculated based on the t-distribution of the log-transformed antibody concentration.
Time Frame: Day 1 (approximately 4 years after completion of the 2+1 schedule)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 177 | 183
EU/mL | 25.99 [21.90 to 30.85] | 2.13 [2.01 to 2.25]

11. Other Pre Specified Outcome: Percentage of Participants With One or More Serious Adverse Events Related to Study Procedure
Description: An SAE is any untoward medical occurrence or effect that at any dose results in death or is life threatening. Life-threatening in this context refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it was more severe.
Time Frame: Up to 4 days following blood sample on Day 1 (approximately 4 years after completion of the 3+1 or 2+1 schedule)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Group Vaxelis (3+1) | Group Infanrix Hexa (3+1) | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Number analyzed (Participants) | 191 | 189 | 181 | 191
Percentage of Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 days after Day 1
Description: Adverse Events (AE) are reported for the Persistence Analysis Set which included all participants previously vaccinated in studies V419-007 or V419-008 with immunogenicity results available. Vaccine safety was not assessed in this study.
Arm/Group | Group Vaxelis (3+1) | Group Infanrix Hexa (3+1) | Group Vaxelis (2+1) | Group Infanrix Hexa (2+1)
Serious Adverse Events (participants affected / at risk) | 0/191 | 0/189 | 0/181 | 0/191
Other Adverse Events (participants affected / at risk) | 0/191 | 0/189 | 0/181 | 0/191

LIMITATIONS AND CAVEATS:
Vaccine safety was not assessed in the present study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations based on these study results 60 calendar days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential will be deleted prior to submission. Whenever needed, Sponsor review may be shorter upon agreement between the Sponsor and the authors.